CLINICAL TRIAL: NCT02500732
Title: A Proof of Principle Study of Atomoxetine for the Prevention of Vasovagal Syncope (VVS): POST6
Brief Title: Prevention of Syncope Trial 6 - Atomoxetine in Vasovagal Syncope
Acronym: POST6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Principal Investigator, Dr. Satish Raj, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POST6; NCT02874937 (obsolete NCT alias)
Record Dates: First submitted 2015-07-13; First posted 2015-07-16 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Vasovagal Syncope
MeSH Terms: conditions — Syncope, Vasovagal | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug was encapsulated in opaque capsules by study personnel not involved in the day to day operations of the study.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule to be given the night before the study tilt, and the morning of the study tilt test.
  Interventions: Drug: Placebo
- Atomoxetine (Active Comparator): Atomoxetine 40mg PO to be given the night before the study tilt, and the morning of the study tilt test.
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — 40mg PO the night before and the morning of the study tilt table test.
  Other Names: Strattera
  Arms: Atomoxetine
Drug: Placebo — oral placebo capsule designed to blind the atomoxetine intervention
  Arms: Placebo

SUMMARY:
Objective: To determine if atomoxetine 40 mg bid (bis in die) in patients ≥18 years old with recurrent vasovagal syncope will better prevent syncope during tilt testing than placebo.

DETAILED DESCRIPTION:
Background: Syncope affects about 50% of Canadians, is the cause of 1-2% of emergency room visits, and probably is responsible for C$250 million (Canadian dollars) in health care spending each year. It is associated with decreased quality of life, trauma, loss of employment, and limitations in daily activities. The most common cause is vasovagal syncope. This occurs in people of all ages, and is a lifelong predilection. While the median number of faints in the population is 2, those who come to the investigators' care have a median 10-15 lifetime spells, and have an increased frequency in the year before presentation. Vasovagal syncope is due to abrupt hypotension and transient bradycardia, which cause cerebral hypoperfusion. The pathophysiology may be either failure of venous return or progressive vasodilation, both due to inappropriately low sympathetic outflow.

There is no known medical treatment for frequent fainting. The investigators performed the pivotal Canadian Institutes of Health Research (CIHR)-funded randomized trials that showed that neither permanent pacing, beta blockers, nor fludrocortisone help the majority of patients. However 2 randomized studies suggest that inhibition of norepinephrine transport (NET) reuptake with sibutramine and reboxetine (NET inhibitors) prevents syncope on tilt testing by about 80%, and the investigators reported that sibutramine markedly reduced the frequency of vasovagal syncope in 7 of our most symptomatic patients. Sibutramine and reboxetine, for different reasons, are not available in Canada. However atomoxetine is available and is used to help patients with attention deficit disorder. There are no data pertaining to its hemodynamic effects in patients with vasovagal syncope. Although a randomized clinical trial of atomoxetine for the prevention of vasovagal syncope would be needed before clinical use, a proof of principle study is needed first.

Objective: To determine if atomoxetine 40 mg bid (bis in die) in patients ≥18 years old with recurrent vasovagal syncope will better prevent syncope during tilt testing than placebo.

Methods: The investigators will conduct a prospective, randomized, parallel, double-blind, proof-of-concept study to test the hypothesis that norepinephrine transporter inhibition with Atomoxetine prevents tilt-induced vasovagal syncope (VVS)/pre-syncope in patients with clinical vasovagal syncope. Subjects will have had ≥1 faint in the previous year, and a diagnosis of vasovagal syncope based on the Calgary Syncope Symptom Score. The primary outcome measure will be the time to syncope or presyncope with a trough rate-pressure product <7000 mm Hg/min. The primary analysis will be performed on an intention-to-treat basis. Secondary analyses will include modelled estimations of systemic vascular resistance and stroke volume, based on arterial waveform and blood pressure. This will permit us to address whether NET inhibition prevents the vasovagal reflex by maintenance of cardiac preload or maintenance of systemic vascular resistance. The investigators will randomize 64 patients in a double blind acute phase 2 study to either Atomoxetine 40mg PO bid x 2 doses or matching placebo.

A sample size of 56 syncope patients would have 85% power to detect a 60% relative risk reduction from a placebo outcome rate of 65%, using an unmatched 2-tailed test with alpha=0.05. To compensate for the report dropout rate we will inflate the sample by 15% to 64 subjects. A formal, blinded mid-way safety and efficacy analysis will be performed with a p<0.01 stopping rule for efficacy. The sample size will be inflated to 74 to account for spending power on the interim analysis. This will provide 85% power to detect an 80% relative risk reduction.

Relevance: This will be the first adequately powered study of the ability of atomoxetine to prevent the vasovagal reflex. It will also provide insight as to whether norepinephrine transport inhibition functions here to maintain venous return or increase systemic vascular resistance. If positive, the study will provide a strong biomedical rationale and preliminary clinical results leading to a randomized clinical trial of atomoxetine for the prevention of vasovagal syncope.

ELIGIBILITY:
Inclusion Criteria:

* 1 or more syncopal spells in the year preceding enrolment
* More than -2 points on the Calgary Syncope Symptom Score
* Age ≥18 years with informed consent

Exclusion Criteria:

* Other causes of syncope, such as ventricular tachycardia, complete heart block, orthostatic hypotension or hypersensitive carotid sinus syndrome
* Inability to give informed consent
* important valvular, coronary, myocardial or conduction abnormality or significant arrhythmia.
* hypertrophic cardiomyopathy
* a permanent pacemaker
* a seizure disorder
* hypertension defined as >150/90 mm Hg
* pregnancy
* glaucoma
* medications with known effects on blood pressure
* Known hypersensitivity to atomoxetine and derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-07; Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Atomoxetine
Started | 27 | 30
Completed | 27 | 29 (Not true event in 1 participant (pseudosyncope))
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atomoxetine | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (14) | 35 (14) | 35 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Calgary Syncope Symptom Score (CSSS) [Median (Full Range); unit: units on a scale] — The Calgary Syncope Symptom Score (CSSS) is a 7-question diagnostic classification scheme that has been validated as a simple point score of historical features, with high sensitivity and specificity for the diagnosis of vasovagal syncope (VVS) in individuals presenting with syncope in the absence of structural heart disease (doi: 10.1093/eurheartj/ehi584). The total CSSS scale ranges from -14 to +6 points. Patients are classified as having tilt-positive primary VVS if the point score is ≥ -2 (i.e. more positive) and syncope due to other causes if the point score is < -2 (i.e. more negative).
  units on a scale | 3 [-2 to 6] | 3 [-2 to 6] | 3 [-2 to 6]
Lifetime Syncope Spells [Median (Inter-Quartile Range); unit: events] | 11 [4 to 20] | 12 [5 to 36] | 12 [5 to 25]
Syncopal Spells in Previous Year [Median (Inter-Quartile Range); unit: events] | 3 [1 to 6] | 3 [2 to 6.75] | 3 [1 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Become Syncopal Associated With Diagnostic Criteria of Hypotension and Bradycardia
Time Frame: 1 hour post start of head up tilt
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 27 | 29
Participants | 19 | 10

2. Secondary Outcome: Number of Participants Who Become Presyncopal (Isolated) Associated With Diagnostic Criteria of Hypotension and Bradycardia
Time Frame: 1 hour post start of head up tilt
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 27 | 29
Participants | 2 | 13

3. Secondary Outcome: Estimated Stroke Volume Index (From the Continuous BP Monitor) During Presyncope
Time Frame: From baseline to within 1 hour post start of head up tilt
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 27 | 29
mL/m2 | 20 (12) | 27 (6)

4. Secondary Outcome: Cardiac Index (From the Continuous BP Monitor) During Presyncope
Time Frame: From baseline to within 1 hour post start of head up tilt
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 27 | 29
L/min/m2 | 1.34 (0.29) | 2.73 (1.10)

5. Secondary Outcome: Systematic Vascular Resistance Index (From the Continuous BP Monitor) During Presyncope
Time Frame: From baseline to within 1 hour post start of head up tilt
Measure: Mean (Standard Deviation); unit: dynes*s/cm5*m2
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 27 | 29
dynes*s/cm5*m2 | 2183 (1238) | 2034 (525)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the week following drug administration.
Arm/Group | Placebo | Atomoxetine
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 0/27 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT02500732/Prot_SAP_000.pdf